CLINICAL TRIAL: NCT04388956
Title: Diagnosis of Thyroid Tumors by Multiple Ultrasonic Factors.
Brief Title: Thyroid Disease Diagnosis by Mutiple Ultrasonic Factors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200805039R
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Thyroid; Nodule; Diagnoses Disease
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months

SUMMARY:
In the outpatient clinic based population setting, the investigators want to reappraise the accuracy of the new model of multi-factorial ultrasound diagnosis with the conventional fine-needle aspiration cytology.

DETAILED DESCRIPTION:
4 to 7 percent of adult population has a palpable thyroid nodule and 17% to 27% of cases can be found when examined by sonography. Although the incidence of the thyroid nodules is high, only 1 of 20 clinically identified nodules is malignant.

Several gray scale sonographic characteristics have been suggestive of malignancy, including hypoechoigenicity, micro calcification, blurred margin and intranodular vascularity. The intranodular vascularity has been studied in several researches. But the previous studies usually evaluated the vascularity by color Doppler sonography and only divided into several categories subjectively. And the result is controversial.

The evaluation of the tumor microcirculation by Doppler ultrasound has been used in many tumors and defined as vascularity index (VI). The power Doppler sonography has many advantages over color Doppler ultrasound in studying the vascularity. It is more sensitive, less noisy. Power Doppler can detect the blood flow of small internal tumor vessels with a diameter of less than 100μm at slow flow rates on the order of a few mm per second1,2 According to our previous study, the vascularity index(PDVI) of thyroid tumor by power Doppler ultrasound between benign and malignant one are statistically different.

In the present study, the investigators examine different PDVI of thyroid tumors and the traditional（B-mode）ultrasound features including the heterogeneity, echogenicity, margin status, and the presence of microcalcification. The investigators consider the several factors simultaneously by statistical model (PCA, FLD). In the outpatient clinic based population setting, the investigators want to reappraise the accuracy of the new model of multi-factorial ultrasound diagnosis with the conventional fine-needle aspiration cytology.

ELIGIBILITY:
Inclusion Criteria:

* patients who have discrete solid thyroid tumors need to undergo fine-needle aspiration cytology to provide the tentative diagnosis
* discrete thyroid tumors with mainly solid content (>50% solid content) and diameter of tumors between 0.5-3cm

Exclusion Criteria:

* abnormal thyroid function, past history of thyroiditis, multinodular goiter, and cystic tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to recruit 300 patients who have discrete solid thyroid tumors need to undergo fine-needle aspiration cytology to provide the tentative diagnosis. The inclusion criteria were discrete thyroid tumors with mainly solid content (>50% solid content) and diameter of tumors between 0.5-3cm. The exclusion criteria were abnormal thyroid function, past history of thyroiditis, multinodular goiter, and cystic tumors.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-07; Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ultrasound evaluation | 3 days
  Patients who were eligible for this trial will receive the new model of ultrasound evaluation . The traditional features including echogenicity, margin, heterogeneity, size and the presence of microcalcification will be recorded in the same time. Then the investigators evaluate the thyroid tumor vascularity in sagittal and transverse section by power Doppler mode (wall filter (WF): medium, colour power angiography (CPA): 82, retroperitoneal fibrosis (RPF): 1000). The DICOM data of the vascularity index(PDVI) will be collected and analyzed later.

CONTACTS AND LOCATIONS:
Overall Officials: Kuen-Yuan Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan